CLINICAL TRIAL: NCT03416907
Title: Informed Consent Formats by Information Preference and Priority
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY2017_00000268
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Consent Forms; Asthma
Keywords: Informed consent
MeSH Terms: conditions — Asthma | interventions — Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Original (Active Comparator): Participants will review the full-length, original consent form for the clinical trial.
  Interventions: Behavioral: Original consent form
- Shortened (Experimental): Participants will review a shortened consent form for the clinical trial, which includes only material indicated as important by 2/3 of participants from a previous study.
  Interventions: Behavioral: Shortened consent form
- Reordered (Experimental): Participants will review a reordered, shortened consent form. This form is based on the shortened consent form, but the sections are reordered based on a previous study, such that sentences previously rated as more likely to impact a participant's decision is more likely to be presented first (except for an initial introductory section).
  Interventions: Behavioral: Reordered, shortened consent form
- Highlighted (Experimental): Participants will review a shortened consent form with a highlights box, where the highlights box includes the 10 sentences rates as most likely to impact a participant's decision from a previous study.
  Interventions: Behavioral: Shortened consent form with a highlights box
- Interactive (Experimental): Participants will review an interactive, shortened consent form, where hyperlinks to different sections of the consent form are provided. The landing page includes the introductory section.
  Interventions: Behavioral: Interactive, shortened consent form

INTERVENTIONS:
Behavioral: Original consent form — Participants will review the full-length, original consent form for the clinical trial.
  Arms: Original
Behavioral: Shortened consent form — Participants will review a shortened consent form for the clinical trial, which includes only material indicated as important by 2/3 of participants from a previous study.
  Arms: Shortened
Behavioral: Reordered, shortened consent form — Participants will review a reordered, shortened consent form. This form is based on the shortened consent form, but the sections are reordered based on a previous study, such that sentences previously rated as more likely to impact a participant's decision is more likely to be presented first (except for an initial introductory section).
  Arms: Reordered
Behavioral: Shortened consent form with a highlights box — Participants will review a shortened consent form with a highlights box, where the highlights box includes the 10 sentences rates as most likely to impact a participant's decision from a previous study.
  Arms: Highlighted
Behavioral: Interactive, shortened consent form — Participants will review an interactive, shortened consent form, where hyperlinks to different sections of the consent form are provided. The landing page includes the introductory section.
  Arms: Interactive

SUMMARY:
This study will test whether different formats of medical informed consent documents can help improve understanding and confidence in decision-making for clinical trials. The study will be primarily run through an online survey.

DETAILED DESCRIPTION:
The goal of this study is to investigate whether the same information can be communicated in different formats of an informed consent document in ways that improve participant understanding and confidence. Participants will review one of several different versions of the same informed consent document, and will be asked to complete a survey after reading the documents. The survey will ask participants their willingness to enroll in the clinical trial discussed in the document and their confidence in their decision. The survey will also test participants recollection of information from the informed consent document. Researchers will look at this data to see if there are ways to improve knowledge about the clinical trial and confidence in decisions without necessarily changing enrollment preferences.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years Old or Older
* Read and agreed to informed consent
* Indicated desire to participate
* Diagnosed with asthma
* US resident

Exclusion Criteria:

* Participants from whom we receive multiple responses will be dropped from analysis (but will be compensated for participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Score for high impact questions | through study completion, an average of 30 minutes
  Sum of correct answers (T/F) for any item relating to material that was rated as 50 or higher on impact on willingness to enroll in a previous study.

SECONDARY OUTCOMES:
Score for low impact questions | through study completion, an average of 30 minutes
  Sum of correct answers (T/F) for any item relating to material that was rated as 49 or lower on impact on willingness to enroll in a previous study.
Total score for all questions | through study completion, an average of 30 minutes
  Sum of correct answers (T/F) on full knowledge test.
Interaction effect of format and importance on likelihood of correct answer | through study completion, an average of 30 minutes
  Interaction effect in a logistic regression predicting a correct answer, based on the format of the consent form and the importance of the answer.
Scores for different information categories | through study completion, an average of 30 minutes
  Sum of correct answers (T/F) for each of the 20 information categories
Effect of location on score | through study completion, an average of 30 minutes
  Logistic regression coefficient of likelihood of predicting a correct answer, based upon the location on which the sentence appeared--uses only the shortened, and the reordered conditions. Note that sentences appearing in the introduction (which is the first section of all treatments) must be dropped, as there will be no variation in location.
Decision to enroll | through study completion, an average of 30 minutes
  Likert measure of participants hypothetical decision to enroll in the study
Confidence in enrollment decision | through study completion, an average of 30 minutes
  Likert measure of participants confidence in hypothetical decision to enroll in the study
Satisfaction with consent structure | through study completion, an average of 30 minutes
  Likert measure of participants satisfaction with the consent form
Perception of investigator concern for well being | through study completion, an average of 30 minutes
  Likert measure of participants belief in the investigator's concerns for the participant's well-being
Perception of investigator transparency | through study completion, an average of 30 minutes
  Likert measure of participants belief that the investigator is trying to communicate information about the trial accurately
Participant's probability estimate of the likelihood that the treatment would help control their asthma | through study completion, an average of 30 minutes
  Survey question of the following form:
  'If you enrolled in the trial described in the consent form, what is the probability that the treatment could help control your asthma better, where 0% means "no chance at all of helping" and 100% means "would definitely help"?'
  Participants provided with drop-down menu including values from 0% to 100% in increments of 1%.

OTHER OUTCOMES:
Participant's free-response text describing what was learned from reading the informed consent document | through study completion, an average of 30 minutes
  Survey question of the following form:
  "What are some of the key things you learned from reading the informed consent document?"
  Participants are then provided with an free-response text box where they are allowed to enter whatever text they want, as long as they enter some text. These responses will be coded by two independent coders, blinded to the treatment arms, using an emergent coding system to identify different topics that participants may raise.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Intend to share deidentified participant data, but we want to review the received data to ensure that there is no information that could potentially reveal individual identity that we may not initially anticipate. As such, a clear delineation of what data will be disclosed is not yet available.